CLINICAL TRIAL: NCT03697525
Title: Effects of Repeated (Focal) Muscle Vibration (rMV) on Motor Recovery After Acute Stroke: a Randomized Sham-controlled Study
Brief Title: Repeated Muscle Vibration in Acute Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Vittorio Di Piero, Associate Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: URomLS - VDiPiero
Record Dates: First submitted 2018-09-29; First posted 2018-10-05 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Acute Stroke
Keywords: repetitive muscle vibration (rMV); acute stroke; motor recovery; nonpharmacological therapy; bedside intervention
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: prospective randomized double-blind sham-controlled study
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vibration Group (VG) (Experimental): VG participants undergo rMV treatment, carried out for three consecutive days by 2 trained physiatrists; each daily session consists of three 10-minute treatment (for each treated limb), interspersed with a 5-minute break. During the rMV, subjects are required to make a voluntary isometric contraction of the treated muscle
  Interventions: Device: Vibration
- Control Group (CG) (Sham Comparator): CG participants undergo the sham rMV by positioning the vibrator close to the tendon but without touching the skin. In this condition, patients were only subject to the faint buzzing sound of the vibrator. Sham rMV treatment is carried out for three consecutive days by 2 trained physiatrists; each daily session consists of three 10-minute treatment (for each treated limb), interspersed with a 5-minute break. During the rMV, subjects are required to make a voluntary isometric contraction of the treated muscle
  Interventions: Device: Vibration

INTERVENTIONS:
Device: Vibration — Low-amplitude rMV (frequency 100 Hz; amplitude range 0.2-0.5 mm) is applied over the flexor carpi radialis and the biceps brachii for the upper limb treatment, and/or over the quadriceps femoris for the lower limb treatment, by means of a specific commercial device (Cro®System, NEMOCOsrl).
  Other Names: Repeated (focal) Muscle Vibration (rMV)

SUMMARY:
prospective randomized double-blind sham-controlled study aimed to investigate the effects of Repeated Muscle Vibration (rMV) on motor recovery in acute stroke patients, treated within 72 hours from symptoms onset

DETAILED DESCRIPTION:
This is a prospective randomized double-blind sham-controlled study. After enrollment (T-0), patients are randomly placed into the vibration group (VG) or the control group (CG), by using a computer-generated randomization list. VG patients receive rMV treatment while those of CG receive the sham one. Both treatments are carried out during the 1st, 2nd and 3rd day after enrollment. Physiokinesitherapy (PT) is carried out in all patients every day, starting soon after T-0 clinical evaluation. Patients are re-evaluated after 4 ± 1 days (T-1), at the end of treatment.

Upon admission, all participants' demographic details and medical history are recorded. All patients undergo a clinical examination, performed at all time-points by an experienced investigator, blinded to group assignment and different from the recruiting one. Clinical evaluation consists of stroke severity evaluation, by means of NIH Stroke Scale; motor and functional limbs abilities are evaluated by using both the Fugl-Meyer scale and the Motricity Index; post-stroke spasticity is assessed with Ashworth scale, modified by Bohannon and Smith.

All participants undergo a daily rehabilitation program. The physical therapist is instructed about duration, frequency, and content of therapy in order to ensure uniformity in treatment procedures, and blinded to patients' treatment allocation.

Low-amplitude rMV (frequency 100 Hz; amplitude range 0.2-0.5 mm) is applied over the flexor carpi radialis and the biceps brachii for the upper limb treatment, and/or over the quadriceps femoris for the lower limb treatment, by means of a specific commercial device (Cro®System, NEMOCOsrl).

The rMV treatment is carried out for three consecutive days by 2 trained physiatrists; each daily session consists of three 10-minute treatment (for each treated limb), interspersed with a 5-minute break.

During the rMV, subjects are required to make a voluntary isometric contraction of the treated muscle.

Otherwise, the CG participants undergo the sham rMV by positioning the vibrator close to the tendon but without touching the skin. In this condition, patients are only subject to the faint buzzing sound of the vibrator

ELIGIBILITY:
Inclusion Criteria:

* age >18,
* first ever stroke detected by Magnetic Resonance Imaging (MRI) or Computer Tomography (CT) scan
* ischemic or hemorrhagic stroke within 72 hours from symptom onset
* motor deficit of the upper and/or lower limb;
* ability to perform at least a minimal isometric voluntary contraction of the affected limb

Exclusion Criteria:

* TIA, or rapidly improving stroke
* cerebral venous thrombosis
* patients presenting with aphasia, neglect, or apraxia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Motor Recovery | 4 ± 1 days
  Motor recovery is expressed as the differences over time (from T-0 to T-1) between the two groups concerning Motricity Index scale scores. The Motricity Index is an ordinal scale that evaluates motor skills and functional limbs in patients with neurological diseases.
  The movements object of the evaluation are in total 6 (3 for each limb) The scores range from 0 (i.e. no movement) to 33 (ie normal movements) for a maximum of 100 for each limb.

SECONDARY OUTCOMES:
Motor Recovery within/associated to synergies | 4 ± 1 days
  Motor recovery occurring within/associated to synergies is expressed as the differences over time (from T-0 to T-1) between the two groups concerning Fugl-Meyer scale scores. This scale consists of 10 subtests (6 subtests for the upper limb and 4 for the lower limbs), which evaluate the movements occurring within the synergies (flexor or extensor) and the movements that occur with the association of synergies.
  It consists of 50 items and provides a maximum score of 100 points, which corresponds to normal traction (66 points for the upper limb, 34 for the lower one) and a minimum score of 0 (no traction)
Stroke Recovery | 4 ± 1 days
  Stroke recovery is expressed as the differences over time (from T-0 to T-1) between the two groups concerning NIH Stroke Scale scores. This scale assesses the stroke severity; it consists of 11 items and the total score goes from a minimum of 0 = normal neurological examination at a maximum of 42, severe severe neurological deficit.
Spasticity Recovery | 4 ± 1 days
  Post-stroke Spasticity is assessed with Ashworth scale, modified by Bohannon and Smith. The total score goes from 0 (no spasticity) to 4 (maximum spasticity grade)

CONTACTS AND LOCATIONS:
Overall Officials: Vittorio Di Piero, Prof, Principal Investigator — Università di Roma La Sapienza
Locations (1):
- Department of Human Neurosciences, "Sapienza" University of Rome, Rome, Italy

IPD SHARING:
Plan to Share IPD: No